CLINICAL TRIAL: NCT04282642
Title: Effects of Computerized Cognitive Brain Training on Sleep, Arousal, and Daytime Functioning in Older Adults With Insomnia
Brief Title: Playing Cognitive Games For Older Adults With Insomnia
Acronym: PLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: American Academy of Sleep Medicine (Other)
Responsible Party: Principal Investigator, Ashley Curtis, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018341
Record Dates: First submitted 2020-02-13; First posted 2020-02-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive training; Sleep; Cognition; Polysomnography; Actigraphy; Older Adults
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the cognitive training or waitlist control(WLC). In both conditions, they will receive the intervention, but the waitlist control will receive this later. Both groups will complete 6 weeks of the cognitive training game either immediately after 1 week baseline (cognitive training group) or after the week 8 assessments (WLC).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Computerized Cognitive Training
  Interventions: Behavioral: Cognitive Training
- WLC (Experimental): Waitlist Control
  Interventions: Behavioral: WLC (Waitlist Control)

INTERVENTIONS:
Behavioral: Cognitive Training — Participants (n=20) provided game console with cognitive training games and activities.
  Arms: Cognitive Training
Behavioral: WLC (Waitlist Control) — Participants (n=20) will receive the cognitive training intervention later, following week 8 assessments.
  Arms: WLC

SUMMARY:
The purpose of this research is to look at the effects of computerized cognitive training on sleep, mental abilities (cognition), and other aspects of daytime functioning, such as mood, and arousal

ELIGIBILITY:
Inclusion Criteria:

* 60+ yrs of age.
* No neurological or psychiatric illness, dementia, or loss of consciousness > 5 mins.
* Nongamers (i.e. <1 hour of video/cognitive training games per week over last 2 years)
* Proficient in English (reading and writing).
* Meet clinical diagnosis for Insomnia.

Insomnia:

* Insomnia complaints for 6+ months.
* Complaints occur despite adequate opportunity and circumstances for sleep.
* Consist of 1+ of the following: difficulty falling asleep, staying asleep, or waking up too early
* Daytime dysfunction (mood, cognitive, social, occupational) due to insomnia.

Exclusion Criteria:.

* Unable to provide informed consent.
* Unable to undergo randomization.
* Cognitive impairments (i.e. mild cognitive impairment, dementia)
* Other sleep disorder (i.e., sleep apnea, Periodic Limb Movement Disorder)
* Severe untreated psychiatric comorbidity that renders randomization unethical
* Using psychotropic or other medications (e.g., beta-blockers) that alter sleep
* Uncorrected visual/auditory impairments
* Participation in nonpharmacological treatment for sleep/fatigue/mood outside the current study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Subjective Cognitive Self-Efficacy- Cognitive Failures Questionnaire | Up to 15 weeks
  A 25-item scale measuring subjective cognition. Participants rate on a scale of 0 (never) to 4 (very often) how often they experience cognitive mistakes and errors in daily tasks.
Objective Cognition- NIH Toolbox Cognitive Battery | Up to 15 weeks
  20-min computerized battery completed in single sitting on iPad.Domains tested include processing speed and attention, visuospatial ability and memory, verbal learning and memory, and executive functioning and working memory.

SECONDARY OUTCOMES:
Objective Behavioral Sleep - Actigraphy | Up to 15 weeks
  Actiwatch 2 (Philips Respironics) is a watch-like device that monitors light and motor activity. Device is worn 24 hours a day for 7 days at each assessment, and during 6 weeks of intervention. Data analyzed by proprietary software using 30s epochs. Validated algorithm will be used to obtain sleep onset latency, wake time after sleep onset.
Circadian Rhythm - Morningness-Eveningness Questionnaire | Up to 15 weeks
  19-item questionnaire that assesses preference for morning, afternoon, and evening activities. Total score reflects degree of "morningness" or "eveningness" type.
Physiological Arousal- Heart Rate Variability | Up to 15 weeks
  Holter monitor assessed 5 min ECG recordings both at rest and during sleep (with PSG).Time index variables: SDNN (standard deviation of normal to normal heartbeat intervals). Spectral index variables: High frequency (0.15-0.4 Hz), low frequency (0.04-0.15 Hz), very low frequency (below 0.04 Hz).
Subjective Arousal-Global Cognitive Arousal-Perceived Stress Scale | Up to 15 weeks
  Perceived Stress Scale is a self-report measure of how life situations are perceived as stressful. The scale consists of 15 items corresponding to everyday situation and participants are asked to rate on a likert scale from 0 (never) to 4 (very often) how often they felt or thought a specific way. Higher scores correspond to higher perceived stress.
Mood- Beck Depression Inventory (II) | Up to 15 weeks
  21-item inventory that asks respondents to rate on a scale of 0 (no depressive feelings) to 3 (most depressive feelings) their feelings towards various aspects of daily living/situations. Higher total scores indicate worse depressive symptoms.
Alcohol Use- Alcohol Use Disorder Test | Baseline
  10-item questionnaire that assess the frequency of alcohol use and problems associated with alcohol use over the past year.
Mood- State-Trait Anxiety Inventory | Up to 15 weeks
  Inventory that asks respondents to rate how true 20 self-descriptive statements (e.g., I feel calm) are on a 4-point scale (1 = not at all, 4 = very much so). Typically, respondents are asked to rate statements according to how they generally feel (trait-anxiety scale) and how they feel in the current moment (state-anxiety scale). Total scores range from 20 to 80, with higher scores indicating greater maladjustment.
Subjective Arousal- Pre-sleep Arousal Scale | Up to 15 weeks
  Pre-sleep Arousal Scale is a 16-item self-report questionnaire comprising both cognitive and somatic manifestations of arousal.
Subjective Arousal- Arousal Predisposition Scale | Up to 15 weeks
  Arousal Predisposition Scale is a 12-item inventory that has been designed to measure the degree to which an individual experiences arousal. Higher scores indicate greater predisposition to arousal.
Subjective Behavioral Sleep- Electronic Daily Sleep Diaries | Up to 15 weeks
  Electronic Daily Sleep Diaries. Online diaries completed each morning (~5 mins) during 1 wk assessment period and 6 weeks of intervention. Diaries measure sleep onset latency, wake time after sleep onset, total sleep time, and sleep quality.
Subjective Behavioral Sleep- Insomnia Severity Index | Up to 15 weeks.
  Brief self-report measure of current perception of insomnia symptom severity, distress and daytime impairment. Commonly used in insomnia treatment outcome research.
Objective Sleep-PSG | Up to 15 weeks
  Single night PSG measured sleep stages.
Game-related experience | Up to 6 weeks
  During the intervention phase for each group, participants will complete "gaming diary" measuring session duration, games played.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Curtis, PhD, Principal Investigator — University of Missouri- School of Medicine
Locations (1):
- University of Missouri, Columbia, Missouri, United States